CLINICAL TRIAL: NCT00523952
Title: A 12-week, Exploratory, Non-comparative, Multi-centre Study to Evaluate the Efficacy and Safety of 0.1% Tacrolimus Ointment Administered in Adults With Moderate to Severe Atopic Dermatitis
Brief Title: Clinical Trial to Assess the Efficacy and Safety of Tacrolimus Ointment Treatment of Atopic Dermatitis in Adult Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FG-506-06-CEE-01
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Dermatitis, Atopic
Keywords: dermatitis, atopic; tacrolimus; adult
MeSH Terms: conditions — Dermatitis, Atopic | interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tacrolimus ointment

INTERVENTIONS:
Drug: tacrolimus ointment — tacrolimus, single arm, 0.1 ointment
  Other Names: Protopic; FK506 Ointment

SUMMARY:
Objective: Assess efficacy and safety of tacrolimus ointment when used in adults with moderate or severe atopic dermatitis. The ointment was applied on the affected skin twice daily for 3 weeks and then once daily until all lesions were cleared

DETAILED DESCRIPTION:
The study was a one arm non-comparative study. The only study medication was Tacrolimus ointment 0.1% (Protopic ® 0.1%).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, any ethnic group, age ≥16
* Moderate to severe atopic dermatitis
* Has given informed consent

Exclusion Criteria:

* Erythroderma
* Pregnant or breast-feeding
* Skin infection on the affected area

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2004-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Rate of patients with at least 50% (i.e. at least moderate) improvement according to the Physician's global evaluation of clinical response between Baseline and the Week 12/End of Study Visit | 12 weeks

SECONDARY OUTCOMES:
Physician's evaluation of clinical response | 12 weeks
Patient's assessment of global response | 12 weeks
Affected body surface area | 12 weeks
Quality of Life at Baseline/Day 1 and Week 12/End of study | 12 weeks
Changes of mEASI | 12 weeks
Incidence of adverse events during the study, including all clinically significant laboratory values | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma GmbH
Locations (25):
- Czechia (7):
  - Brno
  - Hradec Králové
  - Ostrava
  - Pilsen
  - Prague
  - Tábor
  - Ústí nad Labem
- Hungary (6):
  - Budapest
  - Debrecen
  - Győr
  - Kecskemét
  - Miskolc
  - Pécs
- Poland (12):
  - Bialystok
  - Częstochowa
  - Gdansk
  - Katowice
  - Krakow
  - Lodz
  - Lublin
  - Poznan
  - Sopot
  - Szczecin
  - Warsaw
  - Wroclaw